CLINICAL TRIAL: NCT06951620
Title: Optimizing Aerobic Fitness and Functional Response to Exercise in Older Adults
Brief Title: Optimizing Aerobic Fitness in Older Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vermont Medical Center (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Sherrie Khadanga, Principal Investigator, University of Vermont Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: #STUDY00002693; R01AG084636 (NIH)
Record Dates: First submitted 2025-03-13; First posted 2025-04-30 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Aerobic Capacity; High Intensity Interval Training
Keywords: cardiac rehabilitation; HIIT; MICT; exercise in older adults; aerobic capacity

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Patients who recently experienced a myocardial infarction (MI) or percutaneous intervention (PCI; angioplasty, stent placement or valve replacement) and enroll in Phase 2 Cardiac Rehabilitation (CR) may be randomized to High intensity training
  Interventions: Other: HIIT
- Usual Care Group (Experimental): Patients who recently experienced a myocardial infarction (MI) or percutaneous intervention (PCI; angioplasty, stent placement or valve replacement) and enroll in Phase 2 Cardiac Rehabilitation (CR) may be randomized to Moderate intensity training
  Interventions: Other: MICT

INTERVENTIONS:
Other: HIIT — Patients who recently experienced a myocardial infarction (MI) or percutaneous intervention (PCI; angioplasty, stent placement or valve replacement) and enroll in Phase 2 Cardiac Rehabilitation (CR) may be randomized to High intensity training (HIIT)
  Arms: Intervention Group
Other: MICT — Patients who recently experienced a myocardial infarction (MI) or percutaneous intervention (PCI; angioplasty, stent placement or valve replacement) and enroll in Phase 2 Cardiac Rehabilitation (CR) may be randomized to Moderate intensity training
  Arms: Usual Care Group

SUMMARY:
Hospitalization and treatment for cardiovascular disease is one of the main contributors to disability in older adults. Moderate intensity continuous aerobic and resistance training have been the cornerstone of cardiac rehabilitation (CR) for decades to remediate hospital-acquired functional deficits, but some groups receive less or minimal functional benefit from this training. The proposed studies seek to optimize recovery of aerobic fitness and physical function among older cardiac patients using a novel high intensity training regimen with the long-term goal of reducing subsequent disability and improving clinical outcomes.

DETAILED DESCRIPTION:
Clinical events and hospitalization often initiate disability in older adults with cardiovascular disease (CVD) being the primary cause of hospital acquired disability. Cardiac rehabilitation (CR) was designed to correct this disability, with moderate intensity, continuous aerobic training (MICT) as its foundation but some patients, including older adults, receive less functional benefit from MICT. Attention has recently focused on high intensity interval aerobic training (HIIT) as an alternative to MICT because it improves aerobic fitness to a greater extent and is safe and feasible for older adults enrolled in CR; however, neither HIIT nor MICT address age-related atrophy and weakness. Resistance training is a core component of CR meant to correct these deficits, but the moderate intensity resistance training (MIRT) most commonly used has minimal effects on these outcomes. Thus, there is an unmet clinical need for multi-modal exercise interventions that address the unique needs of older adult patients enrolled in CR to optimize improvements in functional recovery and clinical outcomes.

The investigators will conduct the first direct comparison of HIIT+HIRT to MICT+MIRT to improve VO2peak and physical function in older men and women enrolled in CR.

Aim 1: Determine the efficacy of combined HIIT+HIRT vs MICT+MIRT to increase VO2peak in older adult patients enrolled in CR Aim 2: Determine the efficacy of combined HIIT+HIRT vs MICT+MIRT to increase physical function in older adult patients enrolled in CR.

ELIGIBILITY:
Inclusion Criteria:

* >65 years old
* ambulatory
* enrolled in CR at our center following a recent clinical diagnosis of myocardial infarction or percutaneous intervention will be recruited

Exclusion Criteria:

* have an active malignancy (excluding non-melanoma skin cancer or low grade prostate cancer under surveillance)
* unwilling to comply with the exercise prescription they may be assigned to
* have a submaximal performance on entry exercise tolerance test, defined as respiratory exchange ratio <1.0

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 114 (Estimated)
Dates: Start 2025-04-17 (Actual); Primary Completion 2029-03-15 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in Aerobic fitness | Within 4 months of the intake assessment
  Changes in fitness level (peak oxygen uptake) will be measured from intake to completion of the intervention (4 months after intake).
Change in 30 sec sit-to-stand test (STS) | Within 4 months of the intake assessment
  Changes in STS will be measured from intake to completion of the intervention (4 months after intake).

SECONDARY OUTCOMES:
Changes in Quality of Life- Cardiac Specific | Within 4 months of the intake assessment
  Changes in perceived quality of life (MacNew) questionnaires will be measured from intake to completion of the intervention (4 months after intake). The MacNew Heart Disease Health-Related Quality of Life Questionnaire was used. Scores range from 1 to 7, with higher scores indicating better outcomes.
Changes in Depressive Symptoms | Within 4 months of the intake assessment
  Changes in reported depressive symptoms. The Patient Health Questionnaire (PHQ-9) will be measured from intake to completion of the intervention (4 months after intake). Scores range from 0-27 with higher scores associated with severity of depression
Changes in Executive Function (digit span) | Within 4 months of the intake assessment
  Changes in Executive function (digit span) will be measured from intake to completion of the intervention (4 months after intake). The Digit Span subtest of the Wechsler Adult Intelligence Scale-IV (WAIS-IV) was used. Scores range from 1 to 19, with higher scores indicating worse outcomes.
Changes in Executive Function (BRIEF) | Within 4 months of the intake assessment
  Changes in self-reported Executive function problems (BRIEF) will be measured from intake to completion of the intervention (4 months after intake). The Global Executive Composite (GEC) of the Behavior Rating Inventory of Executive Function (BRIEF) was used. T-scores are reported. A T-score of 50 indicates the population mean, and 10 is the standard deviation. Higher T-scores indicate worse outcomes. T-scores above 65 indicate clinically significant problems.
Changes in Executive Function (trail making) | Within 4 months of the intake assessment
  Changes in Executive function (Trail making task) will be measured from intake to completion of the intervention (4 months after intake). The Trail-Making subtest of the Delis-Kaplan Executive Function System (D-KEFS) was used. Scores range from 1 to 19, with higher scores indicating worse outcomes.
Changes in Physical Function (Six Minute Walk Test) | Within 4 months of the intake assessment
  Changes in 6MWT will be measured from intake to completion of the intervention. Distance walked in meters (m) will be recorded.
Changes in Enjoyment of Exercise (PACES) | Within 4 months of the intake assessment
  Changes in Enjoyment of Exercise will be assessed with the validated Physical Activity Enjoyment Scale and will be measured from intake to completion of the intervention. THe score ranges from 0-48 and score below 24 is interpreted as lower enjoyment of physical activity
Changes in Anxiety | Within 4 months of the intake assessment
  Changes in reported anxiety symptoms. The Generalized Anxiety Disorder questionnaire will be measured from intake to completion of the intervention. Rated from 0-7, the higher the score the more anxious

OTHER OUTCOMES:
Maintenance of Fitness Following Intervention | From completion of intervention (4 months) to follow-up (26 weeks).
  Changes in fitness level (peak oxygen uptake) will be measured from intervention completion until follow-up (8 months after intervention completion).

CONTACTS AND LOCATIONS:
Overall Officials: Sherrie Khadanga MD, Principal Investigator, MD, Principal Investigator — University of Vermont Medical Center
Locations (1):
- UVMMC Cardiac Rehabilitation, South Burlington, Vermont, United States

IPD SHARING:
Plan to Share IPD: Undecided